CLINICAL TRIAL: NCT00637156
Title: A Prospective, Randomized, Controlled, Multicenter Pivotal Clinical Trial of the Artificial Cervical Disc-LP at Two Levels for Symptomatic Cervical Disc Disease
Brief Title: Study of the Safety and Effectiveness of the Artificial Cervical Disc - Low Profile Device at Two Adjacent Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESTIGE LP Two Level Study
Record Dates: First submitted 2008-03-03; First posted 2008-03-17 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2017-10

CONDITIONS: Cervical Degenerative Disc Disease; Radiculopathy; Myelopathy
Keywords: Symptomatic DDD at Two Adjacent Levels of cervical spine
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases | interventions — Total Disc Replacement; Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRESTIGE LP Device (Experimental)
  Interventions: Device: PRESTIGE LP device at two adjacent levels
- ATLANTIS Cervical Plate System (Other)
  Interventions: Device: Bi-level fusion with ATLANTIS Cervical Plate System

INTERVENTIONS:
Device: PRESTIGE LP device at two adjacent levels — PRESTIGE LP is a prosthetic device intended to replace a damaged disc in the cervical spine and intended to act as an intervertebral body spacer rather than a fusion device. It is inserted using an anterior surgical approach.
  Other Names: disc; artificial disc; cervical disc
  Arms: PRESTIGE LP Device
Device: Bi-level fusion with ATLANTIS Cervical Plate System — Bi-level anterior cervical fusion procedure involving cortical ring allograft and the ATLANTIS Cervical Plate System.
  Other Names: plate; cervical plate; fusion; cervical fusion
  Arms: ATLANTIS Cervical Plate System

SUMMARY:
The purpose of this clinical investigation is to assess the safety and effectiveness of using the PRESTIGE-LP device in the treatment of patients with symptomatic degenerative disc disease at two adjacent levels of the cervical spine, with overall success being the primary endpoint of the clinical trial. The primary objective is to show non-inferiority of the investigational device to the control treatment. If non-inferiority is established, superiority will also be examined as the secondary objective.

DETAILED DESCRIPTION:
This clinical investigation is being conducted to evaluate the PRESTIGE-LP device's performance at two adjacent cervical levels (C3-C7) in the treatment of patients with symptomatic degenerative disc disease. One-half of the patients in this randomized pivotal clinical trial will be treated at two adjacent cervical levels with the PRESTIGE-LP device. The remaining patients will receive a bi-level anterior cervical discectomy and fusion with cortical ring allografts and the ATLANTIS Cervical Plate System.

ELIGIBILITY:
Inclusion Criteria:

* Has cervical DDD at 2 adjacent cervical levels (C3-C7) requiring surgical treatment & involving intractable radiculopathy, myelopathy, or both
* Has a herniated disc and/or osteophyte formation at each level to be treated that is producing symptomatic nerve root and/or spinal cord compression. The condition is documented by patient history, and the requirement for surgical treatment is evidenced by radiographic studies
* Unresponsive to non-operative treatment for approximately 6 weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management
* Has no previous surgical intervention at the involved levels or any subsequent planned/staged surgical procedure at the involved or adjacent level(s)
* Must be ≥ 18 years; skeletally mature at time of surgery
* Preoperative NDI score ≥ 30
* Preoperative neck pain score ≥ 8 based on the preoperative Neck and Arm Pain Questionnaire
* If a female of childbearing potential, patient is non-pregnant, non-nursing, and agrees not to become pregnant during the study period
* Is willing to comply with the study plan and sign Patient Informed Consent Form

Exclusion Criteria:

* Has a cervical spinal condition other than symptomatic cervical DDD requiring surgical treatment at the involved levels
* Has documented or diagnosed cervical instability relative to adjacent segments at either level, defined by dynamic (flexion/extension) radiographs showing: Sagittal plane translation > 3.5 mm, or Sagittal plane angulation > 20 degrees.
* Has more than two cervical levels requiring surgical treatment
* Has a fused level adjacent to the levels to be treated
* Has severe pathology of the facet joints of the involved vertebral bodies
* Has had previous surgical intervention at either one or both of the involved levels or at adjacent levels
* Has been previously diagnosed with osteopenia or osteomalacia
* Has any of the following that may be associated with a diagnosis of osteoporosis (If "Yes" to any of the below a DEXA Scan will be required to determine eligibility.)

  * Postmenopausal non-Black female over age of 60 who weighs < 140 pounds
  * Postmenopausal female who has sustained a non-traumatic hip, spine, or wrist fracture
  * Male > 70 years
  * Male > 60 years who has sustained a non-traumatic hip or spine fracture
  * If the level of BMD is a T score of -3.5 or lower or a T score of -2.5 or lower with vertebral crush fracture, then the patient is excluded from the study
* Has presence of spinal metastases
* Has overt or active bacterial infection, either local or systemic
* Has insulin dependent diabetes
* Is a tobacco user who does not agree to suspend smoking prior to surgery
* Has chronic or acute renal failure or prior history of renal disease
* Has a documented allergy or intolerance to stainless steel, titanium, or a titanium alloy
* Is mentally incompetent (If questionable, obtain psychiatric consult)
* Is a prisoner
* Is pregnant
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse
* Is involved with current or pending litigation regarding a spinal condition
* Has received drugs that may interfere with bone metabolism within two weeks prior to the planned date of spinal surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs
* Has a history of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers-Danlos Syndrome, or osteogenesis imperfecta)
* Has a condition that requires postoperative medications that interfere with the stability of the implant, such as steroids. (This does not include low-dose aspirin for prophylactic anticoagulation and routine perioperative anti-inflammatory drugs.)
* Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2006-06; Primary Completion 2011-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Burkus, M.D., Principal Investigator — The Hughston Clinic, P.C.
Locations (29):
- United States (29):
  - The Orthopaedic Center; Crestwood Medical Center, Huntsville, Alabama
  - Todd Lanman, MD, FACS, A Professional Corp.;, Beverly Hills, California
  - Bone & Spine Surgery, Colton, California
  - La Jolla Neurological Associates, AMC; Scripps Memorial Hospital La Jolla; Scripps Memorial Hospital Encinitas, La Jolla, California
  - St. Mary's Spine Center; St. Mary's Hospital, San Francisco, California
  - Delaware Neurosurgical Group; Christiana Care Health Systems, Newark, Delaware
  - Spinal Associates, Gulf Coast Hospital, Panama City, Florida
  - Peachtree Neurosurgery, Northside Hospital, Atlanta, Georgia
  - The Hughston Clinic, P.C., Hughston Hospital and Rehabilitation Center, Columbus, Georgia
  - Neuro Spine & Pain Center; Lutheran Hospital, Fort Wayne, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Great Lakes Neurosurgical; Spectrum Health East Campus, Grand Rapids, Michigan
  - Adams Neurosurgery; Mid Michigan Medical Center, Saginaw, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - The Orthopedic Center of St. Louis; Barnes Jewish West County Hospital, Chesterfield, Missouri
  - Montana Neuro Science Institute; St. Patrick's Medical Center, Missoula, Montana
  - University at Buffalo Neurosurgery, Inc. Kaleida Health-Buffalo General Medical center/Gates Vascular Institute, Buffalo, New York
  - Buffalo Neurosurgery Group, West Seneca, New York
  - Crystal Clinic, Inc.; Akron General Medical Center, Akron, Ohio
  - Central Ohio Neurological Surgeons; Mt. Carmel East Hospital, Westerville, Ohio
  - The Center Orthopaedic & Neurosurgical Care & Research, Bend, Oregon
  - OAA Orthopaedic Specialists, Allentown, Pennsylvania
  - Allegheny Neurosurgery; Washington Hospital, Pittsburgh, Pennsylvania
  - Lexington Brain and Spine Institute, West Columbia, South Carolina
  - Center for Sports Medicine and Orthopaedics; Memorial Hospital, Chattanooga, Tennessee
  - East Tennessee Brain & Spine Center, Johnson City Medical Center, Johnson City, Tennessee
  - Central Texas Spine Institute; Health South Surgical Center, Austin, Texas
  - Virginia Brain and Spine; Winchester Medical Center, Winchester, Virginia
  - West Virginia University; Ruby Memorial Hospital, WVU Hospitals, Inc., Morgantown, West Virginia

REFERENCES:
- [Derived] Gornet MF, Lanman TH, Burkus JK, Hodges SD, McConnell JR, Dryer RF, Schranck FW, Copay AG. One-Level Versus 2-Level Treatment With Cervical Disc Arthroplasty or Fusion: Outcomes Up to 7 Years. Int J Spine Surg. 2019 Dec 31;13(6):551-560. doi: 10.14444/6076. eCollection 2019 Dec. PMID 31970051
- [Derived] Gornet MF, Lanman TH, Burkus JK, Dryer RF, McConnell JR, Hodges SD, Schranck FW. Two-level cervical disc arthroplasty versus anterior cervical discectomy and fusion: 10-year outcomes of a prospective, randomized investigational device exemption clinical trial. J Neurosurg Spine. 2019 Jun 21;31(4):508-518. doi: 10.3171/2019.4.SPINE19157. Print 2019 Oct 1. PMID 31226684
- [Derived] Lanman TH, Burkus JK, Dryer RG, Gornet MF, McConnell J, Hodges SD. Long-term clinical and radiographic outcomes of the Prestige LP artificial cervical disc replacement at 2 levels: results from a prospective randomized controlled clinical trial. J Neurosurg Spine. 2017 Jul;27(1):7-19. doi: 10.3171/2016.11.SPINE16746. Epub 2017 Apr 7. PMID 28387616
- [Derived] Gornet MF, Lanman TH, Burkus JK, Hodges SD, McConnell JR, Dryer RF, Copay AG, Nian H, Harrell FE Jr. Cervical disc arthroplasty with the Prestige LP disc versus anterior cervical discectomy and fusion, at 2 levels: results of a prospective, multicenter randomized controlled clinical trial at 24 months. J Neurosurg Spine. 2017 Jun;26(6):653-667. doi: 10.3171/2016.10.SPINE16264. Epub 2017 Mar 17. PMID 28304237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Started | 209 | 188
Completed | 199 | 164
Not Completed | 10 | 24
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System | Total
Number analyzed (Participants) | 209 | 188 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (8.3) | 47.3 (7.7) | 47.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 98 | 215
  Male | 92 | 90 | 182
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 195 | 172 | 367
  Black | 8 | 8 | 16
  Asian | 1 | 3 | 4
  Hispanic | 4 | 4 | 8
  Other | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: inches] | 67.2 (3.9) | 67.6 (4.0) | 67.4 (3.9)
Weight [Mean (Standard Deviation); unit: lbs] | 182.1 (42.6) | 186.3 (37.2) | 184.0 (40.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (5.6) | 28.6 (4.9) | 28.4 (5.3)
Marital Status [Number; unit: participants]
  Single | 25 | 29 | 54
  Married | 146 | 133 | 279
  Divorced | 32 | 23 | 55
  Separated | 4 | 2 | 6
  Widowed | 2 | 1 | 3
Education Level [Number; unit: participants]
  <High school | 21 | 20 | 41
  High school | 63 | 64 | 127
  >High school | 125 | 104 | 229
Worker's Compensation [Number; unit: participants]
  Yes | 26 | 19 | 45
  No | 183 | 169 | 352
Unresolved Spinal litigation [Number; unit: participants]
  Yes | 0 | 1 | 1
  No | 209 | 187 | 396
Alcohol Used [Number; unit: participants]
  Yes | 116 | 88 | 204
  No | 93 | 100 | 193
Preoperative Work Status [Number; unit: participants]
  Yes | 146 | 113 | 259
  No | 63 | 75 | 138

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Success
Description: Rate of overall success is reported as the percentage of participants who met all of the following criteria:
  1. Postoperative Neck Disability Index (NDI) score improvement of at least a 15-point increase from preoperative;
  2. Maintenance or improvement in neurological status;
  3. No serious adverse event classified as implant associated or implant/surgical procedure associated; and
  4. No additional surgical procedure classified as a "failure."
Time Frame: 24 Months
Population: The primary analysis dataset for this study included all subjects who received study devices and completed the initial surgical procedures. The analysis was based on the observed data and missing data due to lost-to-follow-ups were imputed. For the primary endpoint, the analysis consists of 199 investigational subjects and 160 control subjects.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 160
percentage of participants | 81.4 | 69.4
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the overall success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P(p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.113, 95% CI 2-sided [0.022 to 0.201] — The posterior mean of P1-P0, along with the corresponding 95% highest posterior density (HPD) interval, was presented instead of the usual 95% CI
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of overall success rates in two treatment groups was a secondary objective of this trial. Superiority analysis was performed if non-inferiority was demonstrated. If the posterior probability is at least 0.95, a claim of superiority can be made; Test type: Superiority or Other; p = 0.993, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

2. Secondary Outcome: Success Rate of Neck Disability Index
Description: Success rate of Neck Disability Index is reported as the percentage of participants whose neck disability index score met the following criterion: Pre-treatment Score - Post-treatment Score ≥ 15.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable NDI success status at 24 months, which leads to 199 subjects in the investigational group and 159 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 159
percentage of participants | 87.9 | 79.2
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the NDI success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.088, 95% CI 2-sided [0.012 to 0.167] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of NDI success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.990, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

3. Secondary Outcome: Success Rate of Neurological Status
Description: Success rate of neurological status is reported as the percentage of participants who met neurological success defined as maintenance or improvement in all sections (motor, sensory, and reflexes) for the time period evaluated. In order for a section to be considered a success, each element in the section must either remain the same or improve from the time of the preoperative evaluation to the time period evaluated.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable neurological success status at 24 months, which leads to 199 subjects in the investigational group and 159 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 159
percentage of participants | 91.5 | 86.2
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the neurological success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.014 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of neurological success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.931, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

4. Secondary Outcome: Neck Pain Success Rate
Description: Numerical rating scales were used to evaluate pain intensity and frequency. The pain score (0 min, 20 max) was derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and frequency scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Neck pain success rate is reported as the percentage of participants whose neck pain improvement met the following criterion: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable neck pain success status at 24 months, which leads to 199 subjects in the investigational group and 159 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 159
percentage of participants | 98.0 | 95.6
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the neck pain success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.019 to 0.062] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of neck pain success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.852, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

5. Secondary Outcome: Arm Pain Success Rate
Description: Numerical rating scales were used to evaluate pain intensity and frequency. The pain score (0 min, 20 max) was derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and frequency scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Arm pain success rate is reported as the percentage of participants whose arm pain improvement met the following criterion: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable arm pain success status at 24 months, which leads to 199 subjects in the investigational group and 159 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 159
percentage of participants | 88.9 | 89.9
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the arm pain success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 0.997, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = -0.008, 95% CI 2-sided [-0.073 to 0.056] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of arm pain success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.395, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

6. Secondary Outcome: Success Rate of SF-36 PCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success of SF-36 PCS was defined as: Post Score - Pre Score >= 0. The Success rate of SF-36 PCS is reported as the percentage of the participants who were classified as a success for SF-36 PCS.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable SF-36 PCS success status at 24 months, which leads to 197 subjects in the investigational group and 156 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 197 | 156
percentage of participants | 90.4 | 87.8
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the SF-36 PCS success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.024, 95% CI 2-sided [-0.042 to 0.088] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of SF-36 PCS success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.767, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

7. Secondary Outcome: Success Rate of SF-36 MCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success of SF-36 MCS were defined as: Post Score - Pre Score >= 0. The Success rate of SF-36 MCS is reported as the percentage of the participants who were classified as a success for SF-36 MCS.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable SF-36 MCS success status at 24 months, which leads to 197 subjects in the investigational group and 156 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 197 | 156
percentage of participants | 69.0 | 72.4
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the SF-36 MCS success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 0.945, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = -0.024, 95% CI 2-sided [-0.120 to 0.067] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Rate of Disc Height Success
Description: Disc height was assessed by determining the Functional Spinal Unit (FSU) height. The rate of disc height success is reported as the percentage of participants whose disc height for each level based on either the anterior or posterior measurements met the following criterion: Postoperative Height - 6 Week Postoperative Height >= -2mm
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable disc height success (FSU success) status at 24 months, which leads to 170 subjects in the investigational group and 138 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 170 | 138
percentage of participants | 93.5 | 95.7
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the FSU success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 0.997, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = -0.017, 95% CI 2-sided [-0.072 to 0.040] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of FSU success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.271, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

9. Secondary Outcome: Gait Success Rate
Description: Patient's gait was assessed by using Nurick's classification, and indicated either as normal or graded on a scale of 0 to 5. Success was defined as maintenance or improvement in the postoperative status as compared to the preoperative condition: Preoperative Score - Postoperative Score >= 0. The gait success rate is reported as the percentage of participants who had gait success.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable gait success status at 24 months, which leads to 199 subjects in the investigational group and 159 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 199 | 159
percentage of participants | 100.0 | 98.7
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the gait success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.000, Bayesian model — The posterior probability of non-inferiority was calculated and presented instead of the p-value; Risk Difference (RD) = 0.013, 95% CI 2-sided [-0.013 to 0.040] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of gait success rates in two treatment groups was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.859, Bayesian model — The posterior probability of superiority was calculated and presented instead of the p-value

10. Secondary Outcome: Operative Time
Description: Operative time was recorded from skin incision to wound closure.
Time Frame: Time of operation, an average of 1.7-2.1hrs
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
hrs | 2.1 (0.8) | 1.7 (0.7)
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of the operative time in two treatment groups was assessed. The null hypothesis is H0: μ1 = μ0 and the alternative hypothesis is Ha: μ1 ≠ μ0, where μ0 and μ1 denote the mean in control group the investigational group, respectively. Should the posterior probability of superiority P(μ1- μ0 < 0|data) be at least 97.5%, the superiority would be claimed; Test type: Superiority or Other; p = 0.0, Bayesian model — The posterior probably of superiority was calculated and presented instead of the p-value; Posterior Mean Difference = 0.400, 95% CI 2-sided [0.252 to 0.548] — The posterior mean difference (µ1- µ0) and the corresponding 95% highest posterior density (HPD) interval were presented instead of the usual 95% CI

11. Secondary Outcome: Blood Loss
Time Frame: During the time of operation, an average of 1.7-2.1 hrs
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 208 | 188
ml | 67.2 (64.1) | 55.7 (46.3)
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of the blood loss in two treatment groups was assessed.The null hypothesis is H0: μ1 = μ0 and the alternative hypothesis is Ha: μ1 ≠ μ0, where μ0 and μ1 denote the mean in control group the investigational group, respectively. Should the posterior probability of superiority P(μ1- μ0 < 0|data) be at least 97.5%, the superiority would be claimed; Test type: Superiority or Other; p = 0.02, Bayesian model; Posterior Mean Difference = 11.500, 95% CI 2-sided [0.560 to 22.440] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Hospital Stay
Time Frame: From admission to discharge, an average of 1.0-1.5 day
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
days | 1.2 (0.5) | 1.3 (1.0)
Statistical Analysis 1: Comparison: PRESTIGE LP Device vs ATLANTIS Cervical Plate System; Superiority comparison of the hospital stay in two treatment groups was assessed.The null hypothesis is H0: μ1 = μ0 and the alternative hypothesis is Ha: μ1 ≠ μ0, where μ0 and μ1 denote the mean in control group the investigational group, respectively. Should the posterior probability of superiority P(μ1- μ0 < 0|data) be at least 97.5%, the superiority would be claimed; Test type: Superiority or Other; p = 0.892, Bayesian model — The posterior probably of superiority was calculated and presented instead of the p-value; Posterior Mean Difference = -0.100, 95% CI 2-sided [-0.258 to 0.058] — [estimate comment as in outcome 10, analysis 1]

13. Secondary Outcome: Rate of Secondary Surgery at Index Level
Description: Secondary surgical procedures at the index level included revisions, removals, supplemental fixations and reoperations. Rate of secondary surgery at index level is reported as percentage of subjects who had secondary surgeries at index level.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
percentage of participants | 2.4 | 8.0

14. Secondary Outcome: Change of Neck Disability Index Score From Baseline
Description: The self-administered Neck Disability Index (NDI) Questionnaire was used to assess patient neck pain and ability to function. The NDI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability). Change of NDI was defined as NDI at 24 month minus NDI at baseline.
Time Frame: Baseline and 24 months post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
units on a scale
  NDI at baseline (n=209, 188) | 52.1 (13.4) | 53.2 (14.8)
  NDI at 24 months (n=199, 159) | 15.0 (16.6) | 20.0 (20.5)
  NDI change (n=199, 159) | -37.0 (17.8) | -32.5 (19.1)

15. Secondary Outcome: Change of Neck Pain Score From Baseline
Description: Numerical rating scales were used to evaluate neck pain intensity and frequency. Subjects rated their neck pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, subjects recorded their neck pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total neck pain score (0 to 20) was the addition of pain intensity and frequency scores. Change of neck pain score was defined as neck pain score at 24 months minus neck pain score at baseline.
Time Frame: Baseline and 24 months post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
units on a scale
  Neck pain at baseline (n=209, 188) | 16.2 (2.9) | 16.3 (2.6)
  Neck pain at 24 months (n=199, 159) | 4.3 (4.9) | 5.9 (5.5)
  Neck pain change (n=199, 159) | -11.8 (5.2) | -10.3 (5.1)

16. Secondary Outcome: Change of Arm Pain Score From Baseline
Description: Numerical rating scales were also used to evaluate arm pain intensity and frequency. Subjects rated their arm pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, subjects recorded their arm pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total arm pain score (0 to 20) was the addition of pain intensity and frequency scores. Change of arm pain score was defined as arm pain score at 24 months minus arm pain score at baseline.
Time Frame: Baseline and 24 months post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
units on a scale
  Arm pain at baseline (n=209, 188) | 13.8 (5.6) | 14.4 (4.3)
  Arm pain at 24 months (n=199, 159) | 3.0 (4.8) | 4.0 (5.6)
  Arm pain change (n=199, 159) | -10.9 (6.7) | -10.2 (6.5)

17. Secondary Outcome: Change of General Health Status -- SF-36 PCS From Baseline
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS was between 0 and 100, with higher scores denoting better quality of life. Change of SF-36 PCS score was defined as PCS score at 24 months minus PCS score at baseline.
Time Frame: Baseline and 24 months post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
units on a scale
  SF-36 PCS at baseline (n=209, 188) | 31.8 (7.8) | 30.8 (7.4)
  SF-36 PCS at 24 months (n=197, 156) | 47.3 (10.7) | 45.4 (11.5)
  SF-36 PCS change (n=197, 156) | 15.3 (11.5) | 13.8 (11.1)

18. Secondary Outcome: Change of General Health Status -- SF-36 MCS From Baseline
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for MCS was between 0 and 100, with higher scores denoting better quality of life. Change of SF-36 MCS score was defined as MCS score at 24 months minus MCS score at baseline.
Time Frame: Baseline and 24 months post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Number analyzed (Participants) | 209 | 188
units on a scale
  SF-36 MCS at baseline (n=209, 188) | 43.9 (11.8) | 43.8 (12.2)
  SF-36 MCS at 24 months (n=197, 156) | 52.1 (10.8) | 50.9 (10.5)
  SF-36 MCS change (n=197, 156) | 8.1 (14.5) | 6.9 (12.6)

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | PRESTIGE LP Device | ATLANTIS Cervical Plate System
Serious Adverse Events (participants affected / at risk) | 72/209 | 90/188
Other Adverse Events (participants affected / at risk) | 191/209 | 171/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRESTIGE LP Device (N=209) | ATLANTIS Cervical Plate System (N=188)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chronic granulomatous disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Spine malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 7 (7)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abasia (General disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 6 (6) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Device breakage (General disorders) | 0 (0) | 1 (1)
Device connection issue (General disorders) | 0 (0) | 2 (2)
Device dislocation (General disorders) | 3 (3) | 4 (4)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Sensation of pressure (General disorders) | 1 (1) | 0 (0)
Spinal pain (General disorders) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0)
Skin graft infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (4)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cranial nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 10 (11)
Flatback syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Kyphosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 9 (9)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (2) | 0 (0)
Bone scan abnormal (Investigations) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 0 (0) | 1 (1)
Drug screen positive (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Foetal heart rate abnormal (Investigations) | 0 (0) | 1 (1)
Foetal monitoring (Investigations) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neurological examination abnormal (Investigations) | 0 (0) | 1 (1)
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 (1) | 0 (0)
Spinal X-ray abnormal (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
X-ray of pelvis and hip abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (12)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (10)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 11 (12) | 18 (20)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (10)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (12)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (10)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 3 (3)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hypoperfusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 2 (2) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 3 (3) | 2 (2)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 5 (5)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 2 (2)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 2 (2)
Tongue paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Drug dependence (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tobacco user (Social circumstances) | 0 (0) | 1 (1)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric banding (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral nerve decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 2 (2)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 2 (2)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 3 (3)
Vascular stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRESTIGE LP Device (N=209) | ATLANTIS Cervical Plate System (N=188)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Spine malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal cyst (Endocrine disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctival discolouration (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Scintillating scotoma (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 17 (17)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 8 (9)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Adverse drug reaction (General disorders) | 7 (7) | 5 (5)
Asthenia (General disorders) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 6 (6) | 0 (0)
Chest pain (General disorders) | 5 (5) | 3 (3)
Chills (General disorders) | 0 (0) | 2 (2)
Complication of device insertion (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 4 (4)
Device breakage (General disorders) | 1 (1) | 1 (1)
Device connection issue (General disorders) | 0 (0) | 1 (1)
Device deployment issue (General disorders) | 2 (2) | 0 (0)
Device dislocation (General disorders) | 5 (6) | 3 (3)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 2 (2) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Medical device discomfort (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Pain (General disorders) | 12 (12) | 7 (7)
Polyp (General disorders) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 7 (7)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Sensation of foreign body (General disorders) | 1 (1) | 1 (1)
Spinal pain (General disorders) | 1 (1) | 2 (2)
Swelling (General disorders) | 1 (1) | 0 (0)
Tenderness (General disorders) | 1 (1) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 4 (4)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Epidural fibrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 13 (15) | 16 (24)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Heat exhaustion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Inadequate osteointegration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Neck injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve root injury sacral (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 13 (13) | 8 (9)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Angiogram cerebral abnormal (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Biopsy mucosa normal (Investigations) | 1 (1) | 0 (0)
Biopsy oesophagus normal (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 3 (3)
Blood cortisol decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 2 (2)
Blood pressure increased (Investigations) | 3 (3) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Bone scan abnormal (Investigations) | 1 (1) | 1 (1)
Computerised tomogram abnormal (Investigations) | 1 (1) | 0 (0)
False positive investigation result (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1)
Lasegue's test positive (Investigations) | 0 (0) | 1 (1)
Lipids increased (Investigations) | 0 (0) | 1 (1)
Mean cell haemoglobin (Investigations) | 0 (0) | 1 (1)
Neurological examination (Investigations) | 1 (1) | 0 (0)
Neurological examination abnormal (Investigations) | 1 (1) | 3 (3)
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 (0) | 1 (1)
Orthopedic examination abnormal (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Scan abnormal (Investigations) | 1 (1) | 0 (0)
Scan bone marrow abnormal (Investigations) | 1 (1) | 0 (0)
Sensory level abnormal (Investigations) | 0 (0) | 1 (1)
Spinal X-ray abnormal (Investigations) | 0 (0) | 5 (5)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Stress echocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
X-ray abnormal (Investigations) | 0 (0) | 1 (1)
X-ray limb abnormal (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin C deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (21) | 18 (20)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (37) | 35 (39)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cervical spine flattening (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 17 (19) | 11 (13)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (10)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 14 (14) | 12 (12)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 (14) | 19 (24)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 19 (23) | 5 (5)
Joint lock (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 (25) | 12 (16)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 9 (10) | 6 (7)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 (15) | 8 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (11)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 51 (59) | 39 (46)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 16 (18) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 6 (6)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 64 (82) | 60 (77)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (8) | 12 (17)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 (51) | 50 (58)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (7)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal fusion acquired (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 15 (16)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (7)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syndesmophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 10 (13) | 12 (12)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign nipple neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Areflexia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Aura (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 6 (6) | 3 (3)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 11 (11) | 10 (11)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (2) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 3 (3) | 3 (5)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Demyelination (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 2 (2) | 4 (5)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Extensor plantar response (Nervous system disorders) | 0 (0) | 1 (1)
Gait spastic (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Head titubation (Nervous system disorders) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 31 (33) | 35 (44)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 0 (0) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 42 (55) | 38 (47)
Hyporeflexia (Nervous system disorders) | 1 (1) | 4 (5)
Loss of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 2 (2) | 6 (6)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root lesion (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 2 (2)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 33 (42) | 16 (17)
Periodic limb movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Radial nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 2 (2) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis lumbosacral (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3)
Sensory disturbance (Nervous system disorders) | 3 (4) | 2 (2)
Sensory loss (Nervous system disorders) | 6 (6) | 6 (6)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (5) | 0 (0)
Syringomyelia (Nervous system disorders) | 1 (1) | 1 (1)
Tinel's sign (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 4 (4)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1)
Drug dependence (Psychiatric disorders) | 3 (3) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosomatic disease (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Somatoform disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Tension (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Canalith repositioning procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Urostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 7 (7) | 5 (5)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Vasodilatation (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less